CLINICAL TRIAL: NCT06335173
Title: A Phase 2 Double-Blind, Randomized, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Intravenous Sabirnetug in Early Alzheimer's Disease
Brief Title: A Study to Evaluate Efficacy and Safety of Intravenous Sabirnetug in Participants With Early Alzheimer's Disease (ALTITUDE-AD)
Acronym: ALTITUDE-AD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Acumen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACU193-201; 2023-509807-34-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2024-03-13; First posted 2024-03-28 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease
Keywords: Mild Cognitive Impairment; MCI; Mild Alzheimer's Disease; Memory Loss; Memory Problems
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Double-blind Treatment (DBT) Period: sabirnetug 35 mg/kg (Experimental): Participants will receive sabirnetug, 35 milligrams per kilogram (mg/kg), Q4W as intravenous (IV) infusion during the DBT period.
  Interventions: Drug: sabirnetug
- DBT Period: sabirnetug 50 mg/kg (Experimental): Participants will receive sabirnetug, 35 mg/kg, for the first two doses, followed by sabirnetug, 50 mg/kg, Q4W as an IV infusion during the DBT period.
  Interventions: Drug: sabirnetug
- DBT Period: Placebo (Placebo Comparator): Participants will receive sabirnetug matching placebo, Q4W as an IV infusion during the DBT period.
  Interventions: Drug: Placebo
- Open-Label Extension (OLE) Period: sabirnetug 35 mg/kg (Experimental): Participants will receive sabirnetug, 35 mg/kg, Q4W as an IV infusion during the OLE period.
  Interventions: Drug: sabirnetug

INTERVENTIONS:
Drug: sabirnetug — Intravenous sabirnetug
  Arms: DBT Period: sabirnetug 50 mg/kg; Double-blind Treatment (DBT) Period: sabirnetug 35 mg/kg; Open-Label Extension (OLE) Period: sabirnetug 35 mg/kg
Drug: Placebo — Intravenous Placebo
  Arms: DBT Period: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of sabirnetug infusions administered once every four weeks (Q4W) in slowing cognitive and functional decline as compared to placebo in participants with early Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Body weight of at least 30 kilograms (kg) (66 pounds [lbs]) and no more than 160 kg (352 lbs) at Screening
* Must consent to apolipoprotein E4 (APOE4) genotype status assessment
* Must meet all of the following criteria

  1. National Institute on Aging-Alzheimer's Association (NIA-AA) criteria for mild cognitive impairment (MCI) due to Alzheimer's Disease (AD) or probable AD
  2. Screening score between 22 and 30 (inclusive) on the Mini-Mental State Examination (MMSE)
  3. Screening score of 0.5 or 1.0 on the Clinical Dementia Rating Global Score (CDR-GS) and Screening score ≥0.5 on the CDR Memory Box score
  4. Evidence of cerebral amyloid accumulation by either PET scan or CSF
* If using cholinesterase inhibitors or memantine to treat symptoms related to AD, doses must be stable for at least three months (12 weeks) prior to Baseline and every attempt should be made to keep them at stable doses throughout the study
* Must have a reliable informant or study partner who is willing and able to perform all the roles as specified in the study partner Informed Consent Form (ICF)
* Female participants must be surgically sterile or be at least one-year post-menopausal. Male participants with a female partner of child-bearing potential must use adequate contraception

Exclusion Criteria:

* Has any contraindications for MRI studies, including claustrophobia, the presence of metal (ferromagnetic) implants, or a cardiac pacemaker that is not compatible with MRI
* MRI of the brain that is inconsistent with MCI or AD or results showing greater than four ARIA-H, presence of any ARIA-E, or superficial siderosis
* History of significant or unstable neurological disease, other than AD, which may affect cognition or ability to complete the study, such as other dementias, serious infection of the brain, significant head trauma, uncontrolled seizures, stroke, or Parkinson´s disease
* Current serious or unstable clinically important illness that, in the judgment of the site investigator, is likely to affect cognitive assessment including visual and hearing impairment or affect the participant's safety or ability to complete the study
* Malignant disease in the last five years except for resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with a normal posttreatment prostate-specific antibody (PSA)
* Geriatric Depression Scale-Short Form (GDS-SF) score >10 or current symptoms meeting Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V), criteria for major depressive disorder or any current primary psychiatric diagnosis other than AD if, in the judgment of the site investigator, the psychiatric disorder or symptom is likely to confound interpretation of drug effect, affect cognitive assessments, or affect the participant´s ability to complete the study
* Suicide risk, as determined by meeting any of the following criteria:

  1. Any suicide attempt or preparatory acts/behavior on the C-SSRS Baseline/Screening in the last six months
  2. Suicidal ideation in the last six months as defined by a positive response to Question 5 (Suicidal Ideation) on the C-SSRS Baseline/Screening
  3. Significant risk of suicide, as judged by the site investigator
* Conditions that may affect cognitive assessments during the study
* Alcohol use disorder and/or substance use disorder within the last five years

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 542 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Integrated Alzheimer's Disease Rating Scale (iADRS) Score | Baseline up to Week 80
  iADRS is a validated composite of cognition and function made up of Alzheimer's Disease Assessment Scale - Cognitive Subscale 13-item (ADAS-Cog13) and the Alzheimer's Disease Cooperative Study - instrumental Activities of Daily Living scale (ADCS-iADL). ADAS-Cog13 is a rater-administered instrument consisting of 13 items assessing cognitive function areas most typically impaired in AD. ADAS-Cog13 scores range from 0 to 85, with higher scores indicating a greater deficit of global cognition. The ADCS-iADL is a subset of the 23-item ADCS-ADL (items 6a and 7 to 23). The iADLs are more complex skills required to successfully live independently. iADL-items score ranges from 0 to 59 (lower scores indicating greater impairment). The iADRS is calculated as a linear combination of total scores from the ADAS-Cog13 and ADCS-iADL. The iADRS score ranges from 0 to 144 with lower scores indicating worse performance.

SECONDARY OUTCOMES:
Change from Baseline in ADCS-iADL Score | Baseline up to Week 80
  The ADCS-ADL is a 23-item inventory developed as a rater-administered questionnaire to be answered by a participant's study partner, where a participant's performance level is rated over the last 4 weeks, based on a set of performance descriptions. The ADCS-iADL is a subset of the 23-item ADCS-ADL (items 6a and 7 to 23). The iADLs are more complex skills required to successfully live independently, and include shopping, keeping appointments, traveling outside of the home, making a meal or snack, and reading and writing. The iADL-items score ranges from 0 to 59 with lower scores indicating greater impairment.
Change from Baseline in ADAS-Cog13 Score | Baseline up to Week 80
  ADAS-Cog is a rater-administered instrument, designed to assess the severity of dysfunction in cognition, characteristic of persons with AD. The ADAS-Cog13, the cognitive subscale of the ADAS, consists of 13 items assessing cognitive function areas most typically impaired in AD: orientation, verbal memory, language, praxis, delayed free recall, and digit cancellation. The scores range from 0 to 85, with higher scores indicating a greater deficit of global cognition.
Change from Baseline in Clinical Dementia Rating - Sum of Boxes (CDR-SB) | Baseline up to Week 80
  The CDR is obtained through semi-structured interviews of individuals with AD and informants. The ratings are obtained in six domains: memory, orientation, judgment & problem-solving, community affairs, home & hobbies, and personal care. Each domain is rated on a five-point scale of functioning as follows: 0 = no impairment; 0.5 = questionable impairment; 1 = mild impairment; 2 = moderate impairment; and 3 = severe impairment. CDR-SB score is obtained by summing each of the domain scores, with scores ranging from 0 to 18. Higher scores reflect greater cognitive and functional impairment.
Change from Baseline in Mini-Mental State Examination (MMSE) | Baseline up to Week 80
  MMSE is a standard staging and assessment tool in AD, designed for grading the cognitive state of individuals with AD. The scale comprises tasks concerning orientation, memory, attention, language, and praxis to evaluate an individual's cognitive state. MMSE total score ranges from 0 to 30, with lower scores indicative of greater cognitive impairment.
Change from Baseline in Quality of Life in Alzheimer's Disease (QoL-AD) | Baseline up to Week 80
  The QOL-AD tool is a 13-item assessment with each question scored on a 4-point scale where 1 = poor quality of life and 4 = excellent quality of life. Scores range from 13 to 52 with higher scores indicating better quality of life.
Change from Baseline in Neuropsychiatric Inventory Questionnaire (NPI-Q) Score | Baseline up to Week 80
  NPI-Q is a validated questionnaire completed by informants about participants for whom they care. Each of the 12 NPI-Q domains contains a survey question (answered in Yes/No) that reflects the cardinal symptoms of that domain. If the domain response is "Yes," the informant then rates the severity of the symptoms present within the last month on a 3-point scale and the distress of the symptom using a 5-point scale. The total NPI-Q severity score is the sum of the individual severity scores for each symptom and ranges from 0 to 36, with higher scores indicating more severe behavioral impairment. The total NPI-Q distress score is the sum of the individual distress scores for each symptom and ranges from 0 to 60, with higher scores indicating greater caregiver distress.
Change from Baseline in EuroQoL 5-Dimension 5-Level (EQ-5D-5L) | Baseline up to Week 80
  EQ-5D-5L is a self-report survey that measures quality of life. The EQ-5D-5L consists of an EQ-5D descriptive system and EQ visual analog scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels, each assigned a unique 1-digit number: no problems, slight problems, moderate problems, severe problems, and extreme problems. The digits are combined into a 5-digit number that describes the participant's health state. The EQ VAS records the participant's health on a vertical visual analog scale, where the endpoints are labeled 0= the best health you can imagine, and 100= the worst health you can imagine.
Change from Baseline in Resource Utilization in Dementia (RUD) | Baseline up to Week 80
  The RUD questionnaire is a standardized tool and the most widely used instrument for resource use data collection in dementia, enabling comparison of costs of care across countries with differing health care provisions. It is designed to collect data on formal and informal care resource use and to be useful in different care settings, across different countries and care systems, and in both clinical studies and observational cost-of-illness studies.
Change from Baseline in Zarit Burden Interview (ZBI) | Baseline up to Week 80
  ZBI consists of 22 items. Twenty-one of the items are designed to measure several aspects of burden, whereas Item 22 is a global measure of burden. Response options for each item range from 0-4, and total scores range from 0-88, with higher scores indicating greater self-reported burden.
Effect of sabirnetug on Clinical Progression as Compared to Placebo Assessed Using Time Saved Analysis as Measured by iADRS | Baseline up to Week 80
Effect of sabirnetug on Clinical Progression as Compared to Placebo Assessed Using Time Saved Analysis as Measured by ADCS-iADL | Baseline up to Week 80
Effect of sabirnetug on Clinical Progression as Compared to Placebo Assessed Using Time Saved Analysis as Measured by ADAS-Cog13 | Baseline up to Week 80
Effect of sabirnetug on Clinical Progression as Compared to Placebo Assessed Using Time Saved Analysis as Measured by CDR-SB | Baseline up to Week 80
Effect of sabirnetug on Clinical Progression as Compared to Placebo Assessed Using Time Saved Analysis as Measured by MMSE | Baseline up to Week 80
Percentage of Participants with No Clinical Progression at One Year | Baseline up to Week 80
  No clinical progression in participants will be defined as no decline in CDR-SB score. The CDR is obtained through semi-structured interviews of individuals with AD and informants. The ratings are obtained in six domains: memory, orientation, judgment & problem-solving, community affairs, home & hobbies, and personal care. Each domain is rated on a five-point scale of functioning as follows: 0 = no impairment; 0.5 = questionable impairment; 1 = mild impairment; 2 = moderate impairment; and 3 = severe impairment. CDR-SB score is obtained by summing each of the domain scores, with scores ranging from 0 to 18. Higher scores reflect greater cognitive and functional impairment.
Number of Participants with Treatment-Related Adverse Events (TEAEs) | Baseline up to Week 80
Number of Participants with Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI) | Baseline up to Week 80
Number of Participants who Discontinue or Withdraw due to TEAE | Baseline up to Week 80
Number of Participants with Anti-Drug Antibodies (ADA) and Neutralizing Antibodies | Baseline up to Week 80
Number of Participants with Amyloid-Related Imaging Abnormality with Edema/Effusions (ARIA-E) and ARIA with Hemorrhage/Hemosiderin Deposition (ARIA-H) as Measured by Magnetic Resonance Imaging (MRI) | Baseline up to Week 80
Number of Participants with Suicidal Ideation and Behavior as Measured by Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline up to Week 80
  The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe). Greater lethality or potential lethality of suicidal behaviors (endorsed on the behavior subscale) indicates increased risk.
Serum Concentration of sabirnetug | Pre-dose and multiple timepoints post dose up to 80 weeks
Concentration of sabirnetug in Cerebrospinal Fluid (CSF) | Up to Week 76
CSF Concentrations of ACU193 in a Subset of Participants | Up to Week 76
Correlation Between sabirnetug Exposure with Clinical Efficacy Measures | Baseline up to 80 weeks
  Correlation between sabirnetug exposure and clinical outcomes (including iADRS, CDR-SB, ADCS-iADL, ADAS-Cog13, and MMSE) will be assessed in this study.
Change From Baseline in Amyloid Plaque Load or Deposition Measured by Positron Emission Tomography (PET) in Centiloids | Baseline up to Week 76
Change from Baseline in Volumetric Magnetic Resonance Imaging (vMRI) of Whole Brain Volume, Ventricular Volume, and Volume of Selected Regions of Interest | Baseline up to Week 76
Target Engagement Assessed by Measurement of sabirnetug- Amyloid-β oligomer (AβO) Complex in CSF | Up to Week 76
Change from Baseline in CSF Concentrations of Amyloid, Tau and Other Neurodegenerative Biomarkers | Baseline up to Week 76
Change from Baseline in CSF Concentrations of Amyloid, Tau, and Other Neurodegenerative Biomarkers in a Subset of Participants | Baseline up to Week 76
Change from Baseline in Blood Concentrations of Amyloid, Tau, and Other Neurodegenerative Biomarkers | Baseline up to Week 76
Correlation Between Change in Biomarker that Reflect Disease Progression and Clinical Changes | Up to 80 weeks
  Assessment of the correlation between change in clinical outcomes (iADRS, CDR-SB, ADCS-iADL, ADAS-Cog13, and MMSE) and change in biomarker (amyloid PET) will be determined by computing Pearson's correlation coefficient for each treatment group.

CONTACTS AND LOCATIONS:
Locations (68):
- United States (44):
  - The Neurology Center of Southern California - Carlsbad, Carlsbad, California
  - Neurology Center of North Orange County, Fullerton, California
  - Irvine Medical Research, Irvine, California
  - Healthy Brain Research, Long Beach, California
  - Syrentis Clinical Research, Santa Ana, California
  - CenExel - California Neuroscience Research Medical Group, Inc (CNR), Sherman Oaks, California
  - Research Center for Clinical Studies, LLC, Norwalk, Connecticut
  - Re:Cognition Health - Fairfax, Washington D.C., District of Columbia
  - JEM Research Institute, Atlantis, Florida
  - Bradenton Research Center, Bradenton, Florida
  - Gil Fernandez-Yera, MD, PA, Coral Gables, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Coral Clinical Research, Homestead, Florida
  - K2 Medical Research - Villages, Lady Lake, Florida
  - Finlay Medical Research, Miami, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Ocala Health - Family Care Specialists - Ocala I, Ocala, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Alzheimer's Research and Treatment Center - Stuart, Stuart, Florida
  - K2 Medical Research - Tampa, Tampa, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Alzheimers Research and Treatment Center - Wellington, Wellington, Florida
  - Conquest Research, Winter Park, Florida
  - Charter Research - Winter Park, Winter Park, Florida
  - Columbus Memory Center, Columbus, Georgia
  - CenExel - iResearch Atlanta, Decatur, Georgia
  - Office of Jeffrey S. Ross, MD, Northbrook, Illinois
  - Boston Center for Memory, Newton, Massachusetts
  - Hattiesburg Clinic - Memory Center, Hattiesburg, Mississippi
  - ActivMed Practices and Research, Portsmouth, New Hampshire
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - CenExel - Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - Neurological Associates of Albany, Albany, New York
  - AMC Research, Matthews, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Summit Research Network, Portland, Oregon
  - Abington Neurological Associates, Abington, Pennsylvania
  - Keystone Clinical Research, Norristown, Pennsylvania
  - Rhode Island Mood and Memory, East Providence, Rhode Island
  - Neurology Clinic. P.C, Cordova, Tennessee
  - The Alliance for Multispecialty Research LLC (AMR), Knoxville, Tennessee
  - Senior Adult Specialty Research, Austin, Texas
  - Gadolin Research, LLC, Beaumont, Texas
  - Kerwin Medical Center, Dallas, Texas
- Canada (4):
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - Hippocampe d/b/a Ottawa Memory Clinic, Ottawa, Ontario
  - Toronto Memory Program (TMP) (Neurology Research Inc.), Toronto, Ontario
  - MoCA Research and Innovations, Greenfield Park, Quebec
- Germany (4):
  - Charité - Universitaetsmedizin Berlin, Berlin
  - University Hospital of Cologne, Cologne
  - Zentralinstitut für seelische Gesundheit, Mannheim
  - Technical University of Munich, School of Medicine and Health, Klinikum rechts der Isar, Munich
- Spain (8):
  - Hospital Universitari General de catalunya, Sant Cugat del Vallès, Barcelona
  - Fundacion Neuropolis - Hospital Viamed Montecanal, Cuarte de Huerva, Zaragoza
  - Fundacio ACE, Barcelona
  - Policlínica Gipuzkoa, Donostia / San Sebastian
  - Cae Oroitu, Getxo
  - Hospital Ruber, Madrid
  - Hospital Victoria Eugenia, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia
- United Kingdom (8):
  - Re:Cognition Health - London, London, Greater London
  - St. Pancras Clinical Research Ltd., London, Greater London
  - Re:Cognition Health - Winchester, Winchester, Hampshire
  - Neuroclin Glasgow, Motherwell, Lanarkshire
  - Panthera Bio-Partners - Preston, Preston, Lancashire
  - Re:Cognition Health - Guildford, Guildford, Surrey
  - Panthera Biopartners - Sheffield, Sheffield, Yorkshire
  - Re:Cognition Health - Bristol, Bristol

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siemers E, Feaster T, Sethuraman G, Sundell K, Skljarevski V, Cline EN, Zhang H, Jerecic J, Honig LS, Salloway S, Sperling R, Trame MN, Dodds MG, Johnson K. INTERCEPT-AD, a phase 1 study of intravenous sabirnetug in participants with mild cognitive impairment or mild dementia due to Alzheimer's disease. J Prev Alzheimers Dis. 2025 Jan;12(1):100005. doi: 10.1016/j.tjpad.2024.100005. Epub 2025 Jan 1. PMID 39800458